CLINICAL TRIAL: NCT06851650
Title: Early Strengthening of Lower Trapezius and Serratus Anterior Muscles in an Accelerated Rehabilitation Program After Rotator Cuff Repair
Brief Title: Efficacy of Adding Early Scapular Muscles Strengthening Exercise After Rotator Cuff Repair on Scapula Kinematics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Jilan Adel yousef, professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005178
Record Dates: First submitted 2025-02-17; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-09

CONDITIONS: Rotator Cuff Injuries; Rotator Cuff Repair Rehabilition; Supraspinatus Tear
Keywords: Rotator cuff repair Rehabilition, scapular upward rotation, scapular strengthen exercise; accelerate rehabilitation protocol
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early strengthening of Scapular stabilizer muscle and GH Active range of motion (Experimental): Act as study group will receive accelerated protocol with early strengthening of scapular stabilizer muscle of lower trapezius, and serratus anterior and early active GH range of motion (AESA) rehabilitation program.
  Interventions: Other: Rehabilition protocol after rotator cuff repair surgery
- Delay strengthening of Scapular stabilizer muscles and GH Active range of motion (Active Comparator): Act as control group will receive Accelerated protocol with delay strengthening of scapular stabilizer muscles and GH active range of motion (ADSA) rehabilitation program
  Interventions: Other: Rehabilition protocol after rotator cuff repair surgery

INTERVENTIONS:
Other: Rehabilition protocol after rotator cuff repair surgery — adding early scapular strengthening (lower trapezius and serratus anterior) exercise in Rehabilition program after rotator cuff repair surgery

SUMMARY:
The study investigates the effect of accelerate rehabilitation protocol(adding scapular strengthen exercises (lower trapezius and serratus anterior) from week 1) after arthroscopic rotator cuff repair on scapular upward rotation during shoulder elevation.

DETAILED DESCRIPTION:
the study will consist of 2 group Both groups will participate in an accelerated rehabilitation program starting the first week after surgery till week 12, but they will follow different protocols. Accelerated rehabilitation protocol with Early Strengthening of Scapular stabilizer muscle (LT and SA) and GH Active range of motion protocol will be starting gradual active ROM for GH from week 3 post operative till week 12 and gradual scapular muscles strengthening exercises (serratus anterior, lower trapezius) from day 1 while Accelerated rehabilitation protocol with Delay strengthening of Scapular stabilizer muscles and Active GH range of motion protocol will start active ROM for GH and scapular activation exercises (protraction, retraction, and depression) from week 6 till week 12. Patients will wear the sling for the first 6 weeks or as the physician recommends and remove it only during the session and home program.

7 The outcomes will be measured 3 times, at week 3 as a baseline for assessment, then reassess at weeks 6, and 12

ELIGIBILITY:
Inclusion Criteria:

1. Patients after arthroscopic rotator cuff repair.
2. Both gender between age 30 to 50 years
3. Small and medium supraspinatus tear

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Upward rotation of the scapula | At week 3 and week 9 and week 12 after arthroscopic rotator cuff repair
  Measuring the degree of upward rotation of the scapula during shoulder elevation using baseline bubble inclinometer

SECONDARY OUTCOMES:
glenohumeral shoulder elevation | At week 3 and week 9 and week 12 after arthroscopic rotator cuff repair
  Measuring the degree of glenohumeral shoulder elevation using baseline bubble inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- Wengat Hospital, Alexsandria, Egypt

IPD SHARING:
Plan to Share IPD: No